CLINICAL TRIAL: NCT03827265
Title: Transcranial Magnetic Stimulation and Tobacco Use Disorder: A Network-Level Approach With Attention to Sex as a Biological Variable
Brief Title: Transcranial Magnetic Stimulation and Tobacco Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nicole Petersen, Assistant Professor-in-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 18-000509; 1K99DA045749-01 (NIH)
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: This is a single-blind study and only the participant will not be aware of when they will be undergoing the sham stimulation arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- TMS on SFG (Experimental): Device: repetitive transcranial magnetic stimulation (real)
  Transcranial magnetic stimulation (TMS) uses magnetic stimulation to change patterns of activity in your brain. This arm will target the superior frontal gyrus (SFG).
  Other Name: rTMS (active stimulation)
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- TMS on PPC (Experimental): Device: repetitive transcranial magnetic stimulation (rTMS)
  Transcranial magnetic stimulation (TMS) uses magnetic stimulation to change patterns of activity in your brain. This arm will target the posterior parietal cortex (PPC).
  Other Name: rTMS (active stimulation)
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- TMS on dlPFC (Experimental): Device: repetitive transcranial magnetic stimulation (rTMS)
  Transcranial magnetic stimulation (TMS) uses magnetic stimulation to change patterns of activity in your brain. This arm will target the dorsolateral prefrontal cortex (dlPFC).
  Other Name: rTMS (active stimulation)
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- TMS on v5 (Placebo Comparator): Device: repetitive transcranial magnetic stimulation (rTMS)
  Transcranial magnetic stimulation (TMS) uses magnetic stimulation to change patterns of activity in your brain. This arm will target visual cortex (v5).
  Other Name: rTMS (sham stimulation)
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — A rTMS system is an electromagnetic device that non-invasively delivers a rapidly pulsed magnetic field to the cerebral cortex in order to activate neurons within a limited volume without inducing a seizure. The device is intended to be used to treat patients meeting clinical criteria for MDD as defined in the Diagnostic and Statistical Manual of Mental Illnesses, Fourth Edition (DSM-IV). This guidance is issued in conjunction with a Federal Register notice announcing the classification of rTMS systems for the treatment of MDD.

SUMMARY:
The purpose of this study is to determine if brain stimulation using repetitive transcranial magnetic stimulation (rTMS) directed at different parts of the brain can decrease feelings of cigarette craving and symptoms of cigarette withdrawal, and also if men and women have different responses to rTMS.

Participants will visit the University of California, Los Angeles (UCLA) five times: First, for in-person screening, then for four rTMS sessions, four three different brain regions. Everyone in the study will be assigned to all four treatment arms and they will take place in a random order. Before and after each rTMS session, a brief MRI will be performed, and participants will be asked to fill out questionnaires that describe how they are feeling.

DETAILED DESCRIPTION:
After the initial telephone screening, potentially eligible candidates will meet with staff and receive a lay-language explanation of the study. Candidates will review, ask about, and sign the informed consent form for the study. Those who have difficulty understanding the information will be able to review and ask questions to a staff member, who will help clarify the requirements, potential risks and benefits of participation. Any participant who is unable to demonstrate understanding of the information presented despite assistance will be excluded. Participants may withdraw from the study at any time. They may also be withdrawn at the discretion of the investigators for inability to comply with procedures or if continuing participation is unsafe or not in their best interest. Any participant expressing a desire for smoking cessation treatment, at any point during screening or while engaged in the study, will be referred to appropriate counseling services.

Once the informed consent is obtained, participants will undergo a psychological evaluation (MINI) by trained study staff to rule out any exclusionary psychiatric diagnoses. Participants will provide a urine sample to be used for pregnancy and toxicology tests.

They will complete a series of questionnaires to provide demographic information, and complete the Fagerström Test for Nicotine Dependence, Smoking History Questionnaire, Timeline Follow Back (TLFB) to report smoking over the month before testing, Substance Use Inventory, as well as the Beck Depression Inventory, Beck Anxiety Inventory, and Positive and Negative Affect Scale (PANAS) to measure mood state and traits before beginning the study. Daily smoker status will be tested at screening.

Test Day Procedures:

1. Evaluation of wakefulness. Due to the possibility that sleep deprivation may reduce the seizure threshold, wakefulness will be self-reported via the Stanford Sleepiness Scale. Participants who score below a 5 will be asked to reschedule their appointment and return when they are better rested.
2. Abstinence from Drug and Alcohol Use. Each study will begin with a urine test to verify abstinence from drugs of abuse and a Breathalyzer test to verify abstinence from alcohol.
3. Smoking Abstinence. Expired air will be sampled for CO to verify overnight abstinence. Participants who are not abstinent will be allowed to return for testing on another day.
4. Pregnancy Testing. Female participants will each have a urine test to confirm absence of pregnancy.
5. Self-report of Spontaneous Craving. Data will be obtained on the 10-item Urge to Smoke Scale. Self-reports for each item are given on a scale from 1-7, with 1 = definitely not and 7 = definitely.
6. Self-report of Withdrawal. Participants will complete the Shiffman-Jarvik Withdrawal Scale, a 25-item questionnaire comprised of five scales: Craving; Psychological Withdrawal; Physiological Withdrawal; Stimulation/Sedation; and Appetite. Each question is rated on a 7-point scale (1 = definitely not to 7 = definitely) to indicate the respondent's feeling state. Scores are calculated as the mean response to each question on each particular subscale.
7. Self-report of Mood. Participants will complete the Positive and Negative Affect Schedule (PANAS), a 20-item questionnaire comprising two mood scales (positive and negative). Each item is rated on a 5-point scale ranging from 1 (very slightly or not at all) to 5 (extremely) to indicate their feeling state.
8. fMRI. Resting-state fMRI data will be collected while participants lie in the scanner with eyes open viewing a black screen. The scan duration is 8 minutes. Identical scanning procedures will be performed once before rTMS, and once after.
9. rTMS. Subjects will first undergo Motor Threshold (MT) determination using single pulses applied to the left motor cortex, with motor response determined using electromyography (EMG) electrodes applied to the right hand (standard clinical procedures). On active test days, rTMS will be performed using 10 Hz stimulation, a treatment paradigm that has previously reduced craving, with 3000 pulses administered over 15 min at 100% MT with 5 sec pulse trains and 10 sec inter-train interval. Participants will receive this stimulation to the left posterior parietal cortex, dorsolateral prefrontal cortex, and superior frontal gyrus on separate test days.
10. Repeated self-reports of craving, withdrawal, and mood (items 4-6).
11. Repeat fMRI.

Study timeline:

Each of the 4 TMS study visits will be scheduled at least 24 h apart to allow for washout.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Self-identified as male or female
* English fluency;
* Generally good health without cardiovascular, hepatic, renal, or autoimmune diseases; diabetes; or cancer
* Must have smoked for 1 year; smoke 10 cigarettes per day
* Meeting DSM 5 criteria for Tobacco Use Disorder

Exclusion Criteria:

* Seeking treatment for nicotine dependence now or within 3 months before study entry
* A medical condition that may compromise safety
* A neurological disorder that would compromise compliance and/or informed consent
* A major psychiatric disorder
* Current drug use disorders other than Tobacco Use Disorder as defined by DSM 5
* Recent use of drugs of abuse as shown by urine test at the screening or testing sessions
* Smoke marijuana more than once a week
* Use of tobacco in forms other than cigarettes more than 10 days in last month
* Preference for menthol
* Pregnancy or nursing
* Seizure disorder
* Metal implants
* Any other circumstance that the investigators determine would compromise safety

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self-identified as male or female
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Repetitive Transcranial Magnetic Stimulation (rTMS) | 4 weeks
  Data from the brain regions that will be targeted with repetitive transcranial magnetic stimulation (rTMS) will be used to assess changes in craving, withdrawal, and affect
Urge to Smoke Questionnaire | 4 weeks
  A 10-item self-report questionnaire used to measure spontaneous craving
Shiffman-Jarvik Withdrawal Scale | 4 weeks
  A 25-item self-report questionnaire used to measure withdrawal
Positive and Negative Affect Schedule (PANAS) | 4 weeks
  A 20-item questionnaire used to measure mood

SECONDARY OUTCOMES:
Baseline Magnetic Resonance Imaging (MRI) | 4 Weeks
  Resting-state fMRI data will be collected before the TMS session
Post-stimulation Magnetic Resonance Imaging (MRI) | 4 weeks
  Resting-state fMRI data will be collected after the TMS session

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Petersen, Ph.D, Principal Investigator — Faculty
Locations (1):
- Semel Institute of Neuroscience, Los Angeles, California, United States

REFERENCES:
- [Derived] Petersen N, Apostol MR, Jordan T, Ngo TDP, Kearley NW, London ED, Leuchter AF. Comparing neuromodulation targets to reduce cigarette craving and withdrawal: a randomized clinical trial. Neuropsychopharmacology. 2025 Aug;50(9):1319-1326. doi: 10.1038/s41386-025-02106-2. Epub 2025 Apr 25. PMID 40281039